CLINICAL TRIAL: NCT05194150
Title: Performance of Two Non-diffractive Intraocular Lenses With Extended Depth of Vision Set for Mini-monovision
Brief Title: Performance of Two Intraocular Lenses With Extended Depth of Vision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rayner Performance
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cataract Senile
Keywords: Cataract; Cataract surgery; enhanced depth of focus intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rayone EMV (Experimental): Patient will receive the non-diffractive monofocal IOL during cataract surgery
  Interventions: Device: non-diffractive monofocal IOL
- Acrysof IQ Vivity (Experimental): Patient will receive the standard EDOF IOL during cataract surgery
  Interventions: Device: standard EDOF IOL

INTERVENTIONS:
Device: non-diffractive monofocal IOL — Rayone EMV
  Arms: Rayone EMV
Device: standard EDOF IOL — Acrysof IQ Vivity
  Arms: Acrysof IQ Vivity

SUMMARY:
Comparison of the capsular bag performance of two extended depth of vision (EDOF) intraocular lenses (IOLs), the Rayone EMV and the Alcon Acrysof IQ Vivity, in a mini-monovision setting

DETAILED DESCRIPTION:
Spectacle independence is a rising aim in modern cataract surgery. Although bilateral monofocal IOL implantation, aiming for emmetropia leads to high levels of patient satisfaction for distance vision, spectacle dependence for reading and intermediate vision tasks is the usual result.

The option commonly used to achieve spectacle independence in all distances are multifocal intraocular lenses. One concept of multifocality is the trifocal lens. This lens provides good vision in three focal distances: far, intermediate, and near. However, one potential disadvantage of trifocal IOLs is slightly poorer near vision with need for reading gasses for prolonged fine near work and loss of contrast sensitivity in the intermediate distance.

A better intermediate performance concerning contrast vision compared to trifocal IOLs can be reached using enhanced depth of focus (EDOF) lenses. These IOLs have an extended far focus area, which reaches to the intermediate distance, providing high-quality vision over a continuous range of focus, rather than distinct foci with blur in between. In the last years several technologies for EDOF IOLs appeared on the market. The disadvantage compared to monofocal lenses in all of these technologies is the potentially worse contrast sensitivity as well as dysphotopsia.

A new monofocal non-diffractive lens with an extended depth of vision (Rayone EMV) promises an increased range of functional vision and less dysphotopsias. Especially in a monovision setting, where the dominant eye is set for emmetropia and the other eye for low myopia is believe dto be a promising concept for spectacle independence.

Hence, the aim of this study is to compare a new monofocal IOL wit a non-diffractive extended depth of vision (Rayone EMV) with an already established non-diffractive EDOF IOL (Alcon Acrysof IQ Vivity) in a mini-monovision setting.

96 eyes of 48 patients will be included into this study. After randomization, each patient will either receive the Rayone EMV or the Alcon Acrysof IQ Vivity in both eyes. Follow-up visits will be 2 weeks and 3 months after surgery. During these visits a slitlamp examination, measurement of the intraocular pressure, visual acuity assessment, pupil size measurement, determination of the defocus curve, contrast sensitivity measurements, reading speed detection, and a flaremeter measurement will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age-related bilateral cataract
* age 21 or older
* visual acuity > 0.05
* axial length: 22.0 - 26.0 mm
* normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* written informed consent prior to surgery

Exclusion Criteria:

* active ocular disease (e.g. chronic severe uveitis, proliferative diabetic retinopathy, chronic glaucoma not responsive to medication)
* relevant othe rophthalmic diseases such as pseudoexfoliation syndrome (PEX), intraoperative floppy iris syndrome (IFIS)
* corneal decompensation or corneal endothelial cell insufficiency
* previous ocular surgery or trauma
* persons who are pregnant or nursing (pregnancy test will be taken in women of reproductive age)
* corneal astigmatism > 1 dpt.
* retinopathies

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-01-03 (Estimated); Study Completion 2024-01-03 (Estimated)

PRIMARY OUTCOMES:
Visual acuity at intermediate distance | 24 months
  The visual acuity at the intermediate distance will be measured using ETDRS charts at a distance of 80 centimetres and compared between the two different IOLs

SECONDARY OUTCOMES:
Visual acuity at far distance | 24 months
  The visual acuity at the far distance will be measured using ETDRS charts at a distance of 4 metres and compared between the two different IOLs
Visual acuity at near distance | 24 months
  The visual acuity at the near distance will be measured using ETDRS charts at a distance of 40 centimetres and compared between the two different IOLs
Visual acuity in the defocus curve | 24 months
  The visual acuity in the defocus curve will be measured using ETDRS charts at 4 metres with the patient wearing glasses in the power range of -3.5 to +1.0 diopters (presented in 0.5 dioptre steps) and will be compared between the two IOLs
Halometry | 24 months
  The size of the halos depicted in degrees will be assessed using the aston halometer and will be compared between the two IOLs
Contrast sensitivity | 24 months
  Contast sensitvity will be measured using the Optec Vision tester and will be compared between the two IOLs
Reading speed | 24 months
  Reading speed will be assessed with teh Salzburg Reading Desk and will be compared between the two different IOLs

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No